CLINICAL TRIAL: NCT01544673
Title: An Open-label, Placebo-controlled Phase 1 Study to Evaluate the Effect of Linezolid on Ex Vivo Neutrophil and Monocyte Function in Healthy Male Subjects
Brief Title: Effect of Linezolid on Ex Vivo Neutrophil and Monocyte Function in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: A5951164
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Gram Positive Infection
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: linezolid
- Arm B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: linezolid — 600 mg oral tablet twice daily for 4.5 days
  Other Names: Zyvox
  Arms: Arm A
Drug: Placebo — 500 mg oral placebo twice daily for 4.5 days
  Arms: Arm B

SUMMARY:
Results from previous studies have been inconclusive and the effect of linezolid on cytokines remains unclear. This study is designed to evaluate the effect of linezolid on the functionality of white blood cells (neutrophils and monocytes) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 20 and 45 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Subject who had a bacterial/viral infection within 2 weeks prior to the first dose of study medication.
* Subjects with current or prior neutropenia (eg, <1.4 x 109 neutrophils /L).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in phagocytosis of gram-negative bacteria by neutrophils | Baseline, day 4 and day 5
Change from baseline in phagocytosis of gram-negative bacteria by monocytes | Baseline, day 4 and day 5
Change from baseline in interleukin-1 receptor antagonist secretion in response to lipopolysaccharide stimulation | Baseline, day 4 and day 5
Change from baseline in interleukin-1-beta secretion in response to lipopolysaccharide stimulation | Baseline, day 4 and day 5
Change from baseline in interleukin-6 secretion in response to lipopolysaccharide stimulation | Baseline, day 4 and day 5
Change from baseline in interleukin-8 secretion in response to lipopolysaccharide stimulation | Baseline, day 4 and day 5
Change from baseline in tumor necrosis factor alpha secretion in response to lipopolysaccharide stimulation | Baseline, day 4 and day 5

SECONDARY OUTCOMES:
Linezolid peak concentration on day 4 | day 4
Linezolid peak concentration on day 5 | day 5
Linezolid trough concentration on day 5 | day 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951164&StudyName=Effect%20of%20Linezolid%20on%20Ex%20Vivo%20Neutrophil%20and%20Monocyte%20Function%20in%20Healthy%20Males%20